CLINICAL TRIAL: NCT03800420
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled, Phase 2a Study to Evaluate the Efficacy and Safety of BBT-401-1S in Patients With Active Ulcerative Colitis
Brief Title: Efficacy and Safety of BBT-401-1S in Ulcerative Colitis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: to carry out the rest of the study with new CRO and modified protocol as a multi-regional study.
Sponsor: Bridge Biotherapeutics, Inc. (Industry)
Collaborators: KCRN Research, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BBT401-UC-US02
Record Dates: First submitted 2019-01-07; First posted 2019-01-11 (Actual); Results first posted 2022-03-21 (Actual); Last update posted 2022-03-21 (Actual); Status verified 2022-02

CONDITIONS: Ulcerative Colitis
Keywords: Pellino-1
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BBT-401-1S (Experimental): BBT-401-1S, Oral capsule, QD
  Interventions: Drug: BBT-401-1S first and then Placebo
- Placebo (Placebo Comparator): Placebo, Oral capsule, QD
  Interventions: Drug: Placebo first and then BBT-401-1S

INTERVENTIONS:
Drug: BBT-401-1S first and then Placebo — Total 16 week treatment period: The subject takes BBT-401-1S, QD for the first 12 weeks, then placebo for the last 4 weeks.
  Arms: BBT-401-1S
Drug: Placebo first and then BBT-401-1S — Total 16 week treatment period: The subject takes the placebo, QD for the first 8 weeks, then BBT-401-1S for the last 8 weeks.
  Arms: Placebo

SUMMARY:
This is randomized, placebo-controlled, dose-escalation, multicenter, Phase 2 study to evaluate the efficacy and safety of BBT-401-1S in patients with active ulcerative colitis.

This study consists of three cohorts with 16-week treatment period per cohort that will be conducted sequentially.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form (ICF)
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Male or female, aged >=18 years
* Diagnosed with active UC for at least 3 months prior to screening
* Total Mayo score >=5 and Endoscopic sub-score >=1
* Stable dosing regimens of oral drugs (if currently administered) as follows: 5-ASA or sulfasalazine at a stable dose for at least 4 weeks, purine analogues (azathioprine, mercaptopurine, thiopurines) or methotrexate at a stable dose for at least 12 weeks, and low-dose oral corticosteroid (up to 20 mg prednisone/day or equivalent) for at least 4 weeks prior to the first dose of study treatment. Doses of oral drugs must remain stable until the end of study treatment (with possible exception for tapering steroid dose after 8 weeks)
* For females of reproductive potential: use of highly effective contraception for at least 1 month prior to screening and agreement to use such a method during study participation and for an additional 3 months after the last dose
* For males of reproductive potential: use of condoms or other methods to ensure effective contraception with partner during study participation and for an additional 3 months after the last dose

Exclusion Criteria:

* Use of anti-TNF-a biologics or any other biologics for treatment of UC within 60 days prior to randomization.
* Any rectal therapy for treatment of UC or intravenous corticosteroids within 2 weeks prior to randomization.
* Presence of Crohn's disease, indeterminate colitis, ischemic colitis, fulminant colitis, ulcerative proctitis, or toxic mega-colon
* Previous extensive colonic resection (subtotal or total colectomy)
* Ileostomy, colostomy, or known fixed symptomatic stenosis of the intestine
* Evidence of or treatment for Clostridium difficile infection or other pathogenic bowel infection within 60 days or for another intestinal pathogen within 30 days prior to randomization
* Active infection with the HIV or Hepatitis B or C viruses
* Clinically significant active extra-intestinal infection (e.g., pneumonia, pyelonephritis)
* Clinically significant abnormal vital signs, physical examination or 12-lead electrocardiogram (ECG) at screening or baseline
* Clinically significant abnormal results of liver function tests (ALT/AST, bilirubin and alkaline phosphatase) > 2X the upper limit of normal (ULN) at screening
* Other clinically significant abnormal laboratory results at screening in the investigator's opinion
* History of any clinically significant medical condition that, in the investigator's opinion, would preclude participation in the study
* Pregnancy or lactation
* Treatment with another investigational drug or other intervention within 30 days prior to screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2019-04-22 (Actual); Primary Completion 2020-05-18 (Actual); Study Completion 2020-07-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - Site 03, Sacramento, California
  - Site 01, Ventura, California
  - Site 11, Boca Raton, Florida
  - Site 12, Pembroke Pines, Florida
  - Site 04, Rockville, Maryland
  - Site 10, Ann Arbor, Michigan
  - Site 02, Monroe, North Carolina
  - Site 08, Chattanooga, Tennessee
  - Site 05, Austin, Texas
  - Site 13, McAllen, Texas
  - Site 09, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Groups:
- BBT-401-1S: BBT-401-1S, Oral capsule, QD
  BBT-401-1S first and then Placebo: Total 16 week treatment period: Subject takes BBT-401-1S and Placebo. If the subject takes BBT-401-1S, QD for the first 12 weeks, then placebo for the last 4 weeks.
- Placebo: Placebo, Oral capsule, QD
  Placebo first and then BBT-401-1S: Total 16 week treatment period: Subject take BBT-401-1S and Placebo. If the subject takes the placebo, QD for the first 8 weeks, then BBT-401-1S for the last 8 weeks.
Period: Overall Study
Arm/Group | BBT-401-1S | Placebo
Started | 12 | 4
Completed | 10 | 3
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Population: subjects who were randomized
Groups:
- Total: Total of all reporting groups
Arm/Group | BBT-401-1S | Placebo | Total
Number analyzed (Participants) | 12 | 4 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 4 | 15
  >=65 years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 5
  Male | 8 | 3 | 11
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 11 | 4 | 15
  Race: Mixed (White/Black) | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Total Mayo Score
Description: The Total Mayo score is an instrument designed to measure disease activity of ulcerative colitis, with scores ranging from 0 to 12 points. The Total Mayo score consists of 4 subscores( Stool frequency, Rectal bleeding, Findings of endoscopy, Physician global assessment), each graded from 0 to 3 with higher scores indicating more severe disease.
Time Frame: Week 8
Population: No data was collected for this outcome measure due to early termination of study.
Groups:
- BBT-401-1S First and Then Placebo: Total 16 weeks
  First 12 weeks, BBT-401-1S, Oral capsule, QD. Followed by 4 weeks Placebo, Oral capsule, QD.
- Placebo First and Then BBT-401-1S: Total 16 weeks First Placebo, 8 weeks Oral capsule, QD Followed by 8 weeks BBT-401-1S, Oral capsule, QD
Arm/Group | BBT-401-1S First and Then Placebo | Placebo First and Then BBT-401-1S
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Change From Baseline in Partial Mayo Score
Description: The Partial Mayo score is an instrument designed to measure disease activity of ulcerative colitis, with scores ranging from 0 to 9 points. The Partial Mayo score consists of 3 subscores( Stool frequency, Rectal bleeding, Physician global assessment), each graded from 0 to 3 with higher scores indicating more severe disease.
Time Frame: Week 8
Population: No data was collected for this outcome measure due to early termination of study.
Arm/Group | BBT-401-1S | Placebo
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Change From Baseline in Histologic Assessment of Endoscopic Biopsy
Description: Histological assessment of endoscopic biopsy is an appropriate method for evaluating mucosal healing (Carbonnel et al, 1994).
Time Frame: Week 8
Population: No data was collected for this outcome measure due to early termination of study.
Arm/Group | BBT-401-1S | Placebo
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Change From Baseline in Ulcerative Colitis Endoscopic Index of Severity (0-8)
Description: The Ulcerative Colitis Endoscopic Index of Severity (UCEIS) is the first validated index for the assessment of overall endoscopic activity. The model incorporates the vascular pattern score(0-2), the presence of bleeding score(0-3) and the presence of erosions and ulcers score (0-3). Higher score of the sum of these subscore indicates more severe disease.
Time Frame: Week 8
Population: No data was collected for this outcome measure due to early termination of study.
Arm/Group | BBT-401-1S | Placebo
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Number and Severity of TEAEs
Description: Treatment Emergent Adverse Event (TEAE) is defined as an adverse event that occurs or worsens on or after the first dose of study drug.
Time Frame: up to 8 weeks after the last dose
Measure: Number; unit: Number of events
Arm/Group | BBT-401-1S | Placebo
Number analyzed (Participants) | 12 | 4
Number of events
  Abdominal pain | 1 | 0
  Gastrointestinal tract mucosal pigmentation | 1 | 0
  Haemorrhoids | 1 | 0
  Melaena | 1 | 0
  Nasopharyngitis | 1 | 0
  Onychomycosis | 1 | 0
  Condition aggravated | 1 | 0

6. Secondary Outcome: Plasma Concentration of BBT- 401-1S
Description: Analysis of Plasma Pharmacokinetics for BBT- 401 -1S
Time Frame: Day 1, Week 4, Week 8
Population: All samples were below LLOQ and therefore plasma concentrations could not be calculated, (Plasma PK samples of one active patient were not collected.)
Measure: Mean (95% Confidence Interval); unit: ng/ml
Arm/Group | BBT-401-1S | Placebo
Number analyzed (Participants) | 11 | 4
ng/ml | NA [NA to NA] — Samples were below the LLOQ | NA [NA to NA] — Samples were below the LLOQ

7. Secondary Outcome: Change From Baseline in Concentration of Serum CRP
Description: Widely used serum indicator of inflammation in Ulcerative Colitis(UC).
Time Frame: Week 8
Population: No data was collected for this outcome measure due to early termination of study.
Arm/Group | BBT-401-1S | Placebo
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Change From Baseline in Concentration of Fecal Calprotectin
Description: Reliable surrogate marker for disease activity in Ulcerative Colitis (UC).
Time Frame: Week 8
Population: No data was collected for this outcome measure due to early termination of study.
Arm/Group | BBT-401-1S | Placebo
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Change From Baseline in Concentration of Fecal Lactoferrin
Description: A stool (fecal) test that is used to detect inflammation in the intestines.
Time Frame: Week 8
Population: No data was collected for this outcome measure due to early termination of study.
Arm/Group | BBT-401-1S | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 year
Description: TEAEs by MedDRA SOC and PT in study BBT401-UC-US02 . Note 1: A Treatment-Emergent Adverse Event (TEAE) is defined as an adverse event that occurs or worsens on or after the first dose of study drug.
  Note 2: Subjects with one or more adverse events within a level of MedDRA term is counted only once in that level; and percentages are based on the group totals in the column headers.
Arm/Group | BBT-401-1S | Placebo
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/4
Other Adverse Events (participants affected / at risk) | 8/12 | 1/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BBT-401-1S (N=12) | Placebo (N=4)
Colitis ulcerative (Gastrointestinal disorders) | 2 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal tract mucosal pigmentation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Melaena (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 2 (2) | 1 (1)
Onychomycosis (Infections and infestations) | 1 (1) | 0 (0)
Condition aggravated (General disorders) | 1 (1) | 0 (0)
Faecal calprotectin increased (Investigations) | 1 (1) | 0 (0)
Stool analysis abnormal (Investigations) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Institution and Investigator shall not publish the results of this study without the prior written consent of sponsor. As used herein, the term "publish" shall include oral presentations, written abstracts, written manuscripts, etc.

DOCUMENTS (2):
  • Study Protocol (2019-07-19): https://cdn.clinicaltrials.gov/large-docs/20/NCT03800420/Prot_000.pdf
  • Statistical Analysis Plan (2020-07-22): https://cdn.clinicaltrials.gov/large-docs/20/NCT03800420/SAP_001.pdf